CLINICAL TRIAL: NCT03501641
Title: A Study of Heart Rate Variability and Cognitive Load on Image-Based Virtual Reality Instructional Design in Otolaryngology
Brief Title: Heart Rate Variability and Cognitive Load on Image-Based Virtual Reality Instructional Design in Otolaryngology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201601821B0
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Function 1, Social; Competence; Heart Rate Fast; Learning, Spatial; Otolaryngologic Disorder
Keywords: cognitive load; competence; heart rate variation; learning; otolaryngology; video; virtual reality
MeSH Terms: conditions — Tachycardia; Spatial Learning

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will recruit 64 subjects who are novices in otolaryngology at an academic teaching hospital. The cognitive style of the participants is assessed using the Group Embedded Figures Test. The subjects are randomly assigned (1:1) to a novel image-based virtual reality group and conventional video-based group matched by age, sex, and cognitive style.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding to the purpose of the study during recruitment is maintained to minimize preparation bias. After randomization, the participants are unblinded and use image-based virtual reality model or conventional video-based model on a virtual reality eyeglass in an ordinary office environment for 10 minutes. Heart rate variation will be monitored during learning and cognitive load will be assessed by the participants. Subsequently, each participant will perform history taking and physical examination for a real patient in a teaching clinic. The competence will be evaluated using the mini-clinical evaluation exercise, direct observation of procedural skills (DOPS), and milestone assessments. Investigators and outcome assessors are blinded to their randomization and learning models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- image-based virtual reality learning (Experimental): The participants will undergo 10-minute image-based virtual reality learning for history taking and physical examination of otolaryngology.
  Interventions: Other: image-based virtual reality learning
- video-based learning (Active Comparator): The participants will undergo 10-minute video-based learning for history taking and physical examination of otolaryngology.
  Interventions: Other: video-based learning

INTERVENTIONS:
Other: image-based virtual reality learning — The participants will use a whole-view, 360 degree image-based virtual reality to learn a competence of history taking and physical examination for otolaryngology and they can see the response of the staffs and standard patients (including image, voice, face expression, movement, ... etc).
  Arms: image-based virtual reality learning
Other: video-based learning — voice of the staffs and standard patients.
  Arms: video-based learning

SUMMARY:
This study aims to compare heart rate variation, cognitive load, and learning outcomes of novel image-based virtual reality with traditional video in learning for otolaryngology. Half of participants will receive image-based virtual reality learning, while the other half will receive video-based learning.

DETAILED DESCRIPTION:
Background: Workplace-based assessments, such as mini-clinical evaluation exercise (mini-CEX), direct observation of procedural skills (DOPS), and milestones, target the highest level of clinical competence and collect information about doctors' performance in their normal practice. Recent advances in virtual reality (VR) simulation, lowering the complex of learning task and the cognitive load (CL) of the learner, make this novel technology well suited for the initial training of novices. Reduced heart rate variation (HRV), an indicator of stress, is associated with decreased cognitive efficiency in health. Accordingly, this study hypothesizes that VR-based instruction can help novices to increase HRV, decrease CL, and then improve their outcomes of workplace-based assessments.

Aims: This prospective study aims (1) to design an image-based VR (IBVR) instruction for clinical medical education, (2) to compare HRV and CL in traditional video-based (VB) learning and novel IBVR-based learning, (3) to compare outcomes of mini-CEX, DOPS, and milestone between two modules, (4) to perform a qualitative evaluation of IBVR-based learning using a 360-degree video review, and (5) to assess various levels of novice learners (undergraduate medical students and postgraduate year residents) for their participation in and acceptance of this novel IBVR-based learning.

Study Designs: This 3-year study includes two parts: (1) Design a VR-based curriculum including fundamental otolaryngological skills, and (2) Validation of an IBVR-based history taking and physical examination (H&P) learning activity using a blinded randomized, parallel-controlled trial in convenience-sampled novice undergraduate medical students and postgraduate year residents.

Materials and Methods: This study will be implemented between August 1, 2017 and July 30, 2020. Firstly, a VR-based curriculum will be designed including H&P using the analysis, design, development, implementation, and evaluation model and a modified Delphi approach. VB module and IBVR module of the same contexts will be developed. Secondly, an IBVR-based H&P learning activity will be validated by measuring CL questionnaires, reaction time, HRV, mini-CEX, DOPS, milestones, global satisfaction scale and AttrakDiff2 questionnaires (n = 64). Age, sex, and cognitive style (determined by the Group Embedded Figures Test) of both groups are matched. Differences in variables of interests will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 years old;
2. Undergraduate medical students (defined as the last year of medical school training) and postgraduate year residents (defined as the first year after graduation).

Exclusion Criteria:

1. Pregnant, hypertension, recent motion sickness, inner ear infections or claustrophobia, recent surgery, pre-existing binocular vision abnormalities, heart conditions or epileptic symptoms;
2. Declining to participate.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
direct observation of procedural skills (DOPS) | DOPS will be assessed immediately after intervention.
  Procedural skills of history taking and physical examination for otolaryngology will be evaluated using a DOPS assessment immediately after a 10-minute mini-clinical exercise. This assessment uses ten items (indication, explanation, preparation, sites, aseptic/safe procedure, completeness, request for help, recording, interpretation, and global assessment) with 10 (1-10) Likert scales (range: 10-100).

SECONDARY OUTCOMES:
Mini-clinical evaluation exercise (mini-CEX) | The mini-CEX will be assessed immediately after intervention.
  Skills of history taking and physical examination for otolaryngology will be evaluated using a mini-CEX assessment immediately after a mini-clinical exercise. The Mini-CEX is a 10-minute direct observation assessment. This assessment uses seven items (interview, physical examination, professionalism, clinical diagnosis, explanation, efficiency, and global assessment) with 9 (1-9) Likert scales (range: 7-63).
Milestones | The milestones will be assessed immediately after intervention.
  Overall competence of history taking and physical examination for otolaryngology will be immediately evaluated using an assessment of milestones after a 10-minute mini-clinical exercise. This assessment uses five Likert-type levels (basic, focuses, appropriate, accurate, professional) (range: 1-5).
Cognitive Load Scale (CLS) | The CLS will be assessed immediately after intervention.
  Cognitive load of the specific intervention will be immediately evaluated using the Paas CLS questionnaire after an intervention. The Paas CLS questionnaire is a single-item measure of total cognitive load. Participants are asked to rate the perceived intensity of their mental effort with 9 Likert scales (1 = very, very low mental effort; 9 = very, very high mental effort).
Task Load Index (TLX) | The TLX will be assessed immediately after intervention.
  Task Load of the specific intervention will be evaluated using the National Aeronautics and Space Administration TLX questionnaire after an intervention. The questionnaire has six subscales: mental demand; physical demand; temporal demand; performance; effort, and frustration. Participants are asked to indicate the level of each dimension by making a mark on a visual analogue scale with a 21-point Likert scale (range: 0-20). Total cognitive load is interpreted as the sum of the six subscales (range: 0-120).
Cognitive Load Component (CLC) | The CLC will be assessed immediately after intervention.
  Component of cognitive load of the specific intervention will be immediately evaluated using the CLC questionnaire after an intervention. The CLC questionnaire has six subscales: difficulty, complexity, clarity, relevance, focus, and learning with 5 Likert scales (range: 6-30).
Bidirectional feedback and reflection | The bidirectional feedback and reflection will be assessed immediately after intervention.
  Bidirectional feedback and reflection will be immediate evaluated using a qualitative questionnaire after an intervention.
Global Satisfaction Scale (GSS) | The GSS will be assessed immediately after intervention.
  Global satisfaction of the specific intervention will be immediately evaluated using the GSS questionnaire with 11 Likert scales (range: 0-10) after an intervention.
Pragmatic Quality (PQ) | The PQ will be assessed immediately after intervention.
  PQ of the specific intervention will be immediately evaluated using the AttrakDiff2 questionnaire after an intervention. The AttrakDiff2 questionnaire contains 28 questions with 7 Likert-type scales. A PQ scale ranges from -3 to 3.
Hedonic Stimulation (HQ-S) | The HQ-S will be assessed immediately after intervention.
  HQ-S of the specific intervention will be immediately evaluated using the AttrakDiff2 questionnaire after an intervention. The AttrakDiff2 questionnaire contains 28 questions with 7 Likert-type scales. A HQ-S scale ranges from -3 to 3.
Hedonic Identification (HQ-I) | The HQ-I will be assessed immediately after intervention.
  HQ-I of the specific intervention will be immediately evaluated using the AttrakDiff2 questionnaire after an intervention. The AttrakDiff2 questionnaire contains 28 questions with 7 Likert-type scales. A HQ-I scale ranges from -3 to 3.
Attractiveness (ATT) | The ATT will be assessed immediately after intervention.
  ATT of the specific intervention will be immediately evaluated using the AttrakDiff2 questionnaire after an intervention. The AttrakDiff2 questionnaire contains 28 questions with 7 Likert-type scales. A ATT scale ranges from -3 to 3.

OTHER OUTCOMES:
Heart Rate Variation | At baseline for 2 minutes and during an intervention for 10 minutes.
  Before and during an intervention, heart rate is continuously recorded. Heart rate variations will be calculated at baseline and during the specific intervention.
Reaction time | At baseline, the 5th minute and the 10th time.
  The dual-task paradigm with reaction time measurement is manually measured (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ang Lee, MD, MSc, Principal Investigator — Linkou Chang Gung Memorial Hospital, Taoyuan City 33305, Taiwan, ROC
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
No.

REFERENCES:
- [Derived] Lin WN, Chuang HH, Chao YP, Hsin LJ, Kang CJ, Fang TJ, Li HY, Lee LA. Image-based and textbook-based virtual reality training on operational skills among junior residents: a proof of concept study. BMC Med Educ. 2025 May 7;25(1):668. doi: 10.1186/s12909-025-07245-0. PMID 40336062
- [Derived] Chao YP, Chuang HH, Hsin LJ, Kang CJ, Fang TJ, Li HY, Huang CG, Kuo TBJ, Yang CCH, Shyu HY, Wang SL, Shyu LY, Lee LA. Using a 360 degrees Virtual Reality or 2D Video to Learn History Taking and Physical Examination Skills for Undergraduate Medical Students: Pilot Randomized Controlled Trial. JMIR Serious Games. 2021 Nov 22;9(4):e13124. doi: 10.2196/13124. PMID 34813485